CLINICAL TRIAL: NCT06670521
Title: Randomized Trial of Corticosteroids for Post-Extubation Aspiration
Brief Title: Corticosteroids for Post-Extubation Dysphagia
Acronym: COPED
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-1535; R21AG089278 (NIH)
Record Dates: First submitted 2024-09-19; First posted 2024-11-01 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Dysphagia; Laryngeal Edema
MeSH Terms: conditions — Deglutition Disorders; Laryngeal Edema | interventions — Methylprednisolone; Saline Solution

STUDY DESIGN:
Intervention Model Description: Multicenter prospective randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticosteroid Intervention (Experimental): 50 mg Methylprednisolone IV every 6 hours for 4 doses (total dose 200mg)
  Interventions: Drug: Methylprednisolone
- Placebo Control (Placebo Comparator): Normal Saline placebo dose IV every 6 hours for 4 doses
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Methylprednisolone — 50 mg methylprednisolone IV every 6 hours for 4 doses to reduce laryngeal edema
  Arms: Corticosteroid Intervention
Drug: Normal Saline — Normal Saline placebo IV every 6 hours for 4 doses
  Arms: Placebo Control

SUMMARY:
This is a placebo-controlled, double-blind randomized trial of a short course of intravenous corticosteroids for Acute Respiratory Failure Survivors with Fiberoptic Endoscopic Evaluation of Swallowing (FEES) documented laryngeal edema. Study was leveraged using the existing R01 grant infrastructure COMIRB # 21-3873, study design, and research methods. Patients for the study proposed will have already been enrolled in the R01 longitudinal cohort study. The sites to perform this study include Colorado, BU, Yale, and Stanford. Those R01-enrolled patients with laryngeal edema on their initial FEES examination: defined as the revised Patterson edema score greater than zero, will be approached for enrollment.

DETAILED DESCRIPTION:
This is a multicenter study conducted across the University of Colorado, Boston University, Stanford University, and Yale University. The study aims to enroll a total of 80 participants, with approximately 20 participants at each site. This study aims to investigate the effects of intravenous corticosteroids on laryngeal edema and swallowing function in survivors of acute respiratory failure (ARF) who have documented laryngeal edema. It evaluates whether administering corticosteroids can reduce edema and improve quality of life related to swallowing after hospital discharge. The study includes ARF survivors with confirmed laryngeal edema, who will be randomized into two groups. Patients in the intervention group will receive 50 mg of methylprednisolone intravenously every six hours for a total of four doses, amounting to 200 mg (equivalent to 1,000 mg of hydrocortisone), while the control group will receive a saline placebo intravenously under the same regimen.

The primary outcomes of the study focus on measuring the reduction in laryngeal edema post-treatment and evaluating post-extubation swallowing function. Secondary outcomes include assessing quality of life one month after hospitalization, particularly regarding swallowing function and the ability to return to pre-hospitalization dietary habits. To measure laryngeal edema, the Revised Patterson Edema Scale will be utilized, which assesses edema across eight specific regions of the upper airway (such as the epiglottis and vallecula). Each area is rated on a scale from 0 to 3, resulting in an overall score ranging from 0 (normal) to 24 (severe edema). This scale has been adapted for the study to enhance sensitivity and reliability, showing moderate to good interrater reliability across assessed areas.

Participants will be randomized in a 1:1 ratio using a permuted block randomization method to ensure balanced allocation. The findings from this study could have significant implications for post-extubation care in ARF survivors, potentially guiding clinical practices for managing laryngeal edema and improving patients' swallowing function and overall quality of life after hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Participant enrolled in primary study COMIRB #21-3873/ NCT # 05108896
* Laryngeal edema identified on participants primary study Fiberoptic Endoscopic Evaluation of Swallowing (FEES) as defined as a revised Patterson edema score greater than zero
* Admission to an ICU during their hospitalization
* Mechanical ventilation with an endotracheal tube for greater than 48 hours.
* Extubation except for compassionate extubation or transition to end-of-life care.

Exclusion Criteria:

* Patient or provider refusal
* Contraindication or corticosteroids defined as an allergic reaction (extremely rate) or taking other immunosuppressive medications.
* Chronic treatment with corticosteroids (>= 40 mg Prednisone/day, >=32 Methylprednisolone/day)
* Contraindication to enteral/oral nutrition administration.
* Pre-existing history of dysphagia or aspiration.
* Pre-existing or acute primary central or peripheral neuromuscular disorder.
* Presence of a chronic tracheostomy (present prior to ICU admission).
* Pre-existing head and neck cancer or surgery.
* Coagulopathy resulting in uncontrolled nasal or pharyngeal bleeding.
* Delirium as assessed by CAM-ICU
* Inability to obtain informed consent from patient or an appropriate surrogate.
* Age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Pre/post intervention change in the revised Patterson edema scale on FEES exam | Day 1 through Day 5
  Investigators hypothesize that corticosteroids will be more effective (a larger pre/post reduction in the revised Patterson Edema scale) for resolution of swallowing dysfunction in patients recovering from acute respiratory failure with the presence of laryngeal edema on a FEES examination. Change is defined as the pre-study total FEES revised Patterson Edema scale minus the post-study total FEES revised Patterson Edema scale. Improvement in the total revised Patterson Edema scale would a positive number. For example, the pre-study total score was 15, the post-study total score was 8; therefore, the change would be a score of 7. Improvement in the total revised Patterson Edema scale would a positive number

SECONDARY OUTCOMES:
Change in Individual Components of the Revised Patterson Edema Scale | Day 1 through Day 5
  Since there is variability in the amount of edema in the eight different locations of the revised Patterson edema scale, investigators will examine the effect of corticosteroids compared to placebo on the change in edema in each of these eight areas. Change is defined as the pre-study FEES revised Patterson Edema scale minus the post-study FEES revised Patterson Edema scale. The scale assesses eight areas of the upper airway (epiglottis, vallecula, pharyngoepiglottic folds, aryepiglottic folds, arytenoids, false vocal cords, true vocal cords, and pyriform sinuses) using a normal, mild, moderate, or severe scale. For this proposal, we have adapted this rating system to a 0-3 scale (normal =0 and severe = 3) for each of the eight locations in the upper airway. The overall score can range from 0 (normal) to 24 (severe edema in all 8 areas). The overall interrater reliability of the revised Patterson scale maintains moderate-good agreement for each of the eight upper airway locations.
Change in the Penetration-Aspiration Scale (PAS) Score | Day 1 through Day 5
  Investigators will determine whether the administration of corticosteroids results in improvement in the severity of dysphagia and aspiration. The PAS score is a validated measure of the degree of aspiration on FEES of the visualized swallowed bolus. A PAS score of 2-5 defined penetration of the bolus into the laryngeal area above the vocal cords but without entering the airway. A PAS score of 6 or greater defines as aspiration. A PAS score of 6-7 represents non-silent aspiration, and a score of 8 represents silent aspiration. Investigators will determine a PAS score for each bolus during the two FEES examinations.

OTHER OUTCOMES:
Return to Pre-Hospitalization Diet | 1 month post-hospital discharge
  Participants will be contacted by telephone one month after hospital discharge to assess their return to Pre-Hospitalization Diet. A pre-hospitalization diet has already been established in the primary study, 21-3873. Study personnel will ask participants about their current diet post-discharge. Returning to the pre-hospitalization diet will be defined as resuming the same diet they followed before hospitalization.
Post-Discharge Eating Assessment Tool (EAT-10) | 1 month post-hospital discharge
  Participants will be contacted by telephone one month after hospital discharge to complete dysphagia screening tool to identify people at high risk of swallowing disorders. Each item corresponds to 5 difficulty levels from "no problem" to "serious problem," with a total score of 0 to 40. EAT-10 has good internal consistency and intraclass correlation coefficients (ICCs).
Post-Discharge Positive and Negative Affect Schedule (PANAS-SF) | 1 month post-hospital discharge
  Participants will be contacted by telephone one month after hospital discharge to complete 20-item questionnaire to assess positive affect (PA) and negative affect (NA). PA is associated with pleasurable engagement with the environment, whereas NA reflects a dimension of general distress summarizing a variety of negative states such as anger, guilt, or anxiety.
  Positive Affect Score: Add the scores on items 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19. Scores can range from 10 - 50, with higher scores representing higher levels of positive affect. Mean Scores: 33.3 (SD±7.2) Negative Affect Score: Add the scores on items 2, 4, 6, 7, 8, 11, 13, 15, 18, and 20. Scores can range from 10 - 50, with lower scores representing lower levels of negative affect. Mean Score: 17.4 (SD ± 6.2)
Post-Discharge Caregiver Assistance Scale (CAS) | 1 month post-hospital discharge
  Participants will be contacted by telephone one month after hospital discharge to complete an assessment tool to collect data on how much assistance the caregiver provides to the participant for various activities over the past month. A rating of zero (0) indicates "no" assistance is provided, while a rating of six (6) indicates "a lot" is provided.
Post-Discharge Caregiving Impact Scale (CIS) | 1 month post-hospital discharge
  Participants will be contacted by telephone one month after hospital discharge to complete an assessment tool to measure how much the participant's caregiver responsibilities interfere with different aspects of their life in their current living situation. Scoring ranges from zero (0), "Not at all" to six (6), "Very Much". If an item is not applicable, please circle zero (0) to indicate this.
Post-Discharge 20-Item Medical Outcomes Study (MOS) Social Support Survey | 1 month post-hospital discharge
  Participants will be contacted by telephone one month after hospital discharge to complete this survey to measure the availability of support for the participant in several domains. The survey comprises of 4 subscales and one overall summary index. The subscales include emotional/informational support, tangible support, affectionate support, and positive social interaction. The summary score is the overall social support. Scoring ranges from (1) "None of the time to" (6) "All of the time" for each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Moss, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No